CLINICAL TRIAL: NCT06800859
Title: Establishment of a Predictive Model for Post-dural Puncture Headache
Status: Enrolling by invitation | Type: Observational
Sponsor: Yilin Zhao (Other)
Responsible Party: Sponsor-Investigator, Yilin Zhao, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 101787
Record Dates: First submitted 2025-01-17; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Spinal and Epidural Anaesthesia-Induced Headache During Pregnancy
Keywords: Spinal anestheisa; Pural-Puncture; Headache; Complications
MeSH Terms: conditions — Headache | interventions — Bed Rest; Blood Patch, Epidural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- No Post-dural Puncture Headache Group in adult: Perform MRI and (or) ultrasound and (or) intraocular pressure measurement before and 24 hours after the puncture
- Post-dural Puncture Headache Group in adult: Perform MRI and (or) ultrasound and (or) intraocular pressure measurement before and 24 hours after the puncture
  Interventions: Drug: Supplement fluids
- No Post-dural Puncture Headache Group in children: Perform MRI and (or) ultrasound and (or) intraocular pressure measurement before and 24 hours after the puncture
- Post-dural Puncture Headache Group in children: Perform MRI and (or) ultrasound and (or) intraocular pressure measurement before and 24 hours after the puncture
  Interventions: Drug: Supplement fluids

INTERVENTIONS:
Drug: Supplement fluids — To ensure optimal recovery and manage potential complications, patients are advised to supplement fluids by increasing their oral intake or receiving intravenous fluids as necessary. Bed rest is recommended to reduce physical strain and promote healing. Additionally, a blood patch procedure may be performed to alleviate symptoms such as headaches that can occur after certain medical procedures, particularly spinal taps. This involves injecting a small amount of the patient's own blood into the epidural space to seal any leaks of cerebrospinal fluid, thereby providing relief and aiding in recovery. Proper monitoring and follow-up care are essential to ensure the effectiveness of these interventions
  Other Names: Bed rest; Blood patch
  Groups: Post-dural Puncture Headache Group in adult; Post-dural Puncture Headache Group in children

SUMMARY:
The goal of this clinical trial is to establish a predictive model for post-dural puncture headache. The main questions it aims to answer are:

Changes in intracranial pressure after spinal puncture (or lumbar puncture). When post-dural puncture headache occurs, the optic nerve sheath diameter (ONSD) change When the optic nerve sheath diameter (ONSD) and (or) Intraocular Pressure (IOP) reaches a certain threshold, does proactive treatment reduce the incidence of postoperative headaches? Researchers will measure the optic nerve sheath diameter (ONSD) using ultrasound and ( or ) magnetic resonance imaging (MRI) before and after spinal puncture.

Researchers will measure the Intraocular Pressure (IOP) using ICARE before and after spinal puncture.

Participants will:

Undergo ultrasound and (or) magnetic resonance imaging (MRI) examinations before and after spinal puncture Undergo ICARE examinations before and after spinal puncture

DETAILED DESCRIPTION:
Post-dural Puncture Headache (PDPH) refers to a specific type of headache that occurs after patients receive intrathecal anesthesia or a lumbar puncture, resulting from the leakage of cerebrospinal fluid (CSF) due to the puncture of the dura mater and arachnoid mater. This type of headache typically occurs within 24 to 48 hours after the puncture and is characterized primarily by positional headaches, meaning that the headache worsens when the patient is standing or sitting and improves when lying down. The headache is often accompanied by symptoms such as neck stiffness, nausea, vomiting, tinnitus, and blurred vision.

The primary mechanism of PDPH is the leakage of cerebrospinal fluid from the puncture site after the dura and arachnoid are punctured, leading to a decrease in CSF pressure. The reduction in cerebrospinal fluid can cause several physiological changes:Decreased CSF Pressure: The reduction of CSF leads to a drop in intracranial pressure, which alters the mechanisms that support the brain, resulting in pain.Meningeal Tension: The decrease in CSF may cause tension on the meninges and nerve roots, leading to pain sensations.Vasodilation: The drop in intracranial pressure can trigger a reflexive dilation of cerebral blood vessels, further exacerbating the pain.The incidence of PDPH is associated with various factors, including the patient's age, sex, body type, type of surgery performed, and the type and size of the puncture needle used. Smaller needles (such as 25G or thinner) and non-cutting needles (such as Sprotte needles) can significantly reduce the incidence of PDPH, whereas larger and cutting needles (such as Quincke needles) are associated with a higher incidence. Younger patients and females are more prone to developing PDPH. Additionally, multiple punctures increase the risk of PDPH.

Timely and effective treatment can significantly reduce the occurrence of PDPH; however, there is currently a lack of monitoring methods for PDPH. This study aims to establish a predictive model for the occurrence of PDPH by measuring postural cerebrospinal fluid pressure using ultrasound, which can enable early prediction and treatment of PDPH, thereby significantly improving patient comfort and recovery processes.

The goal of this clinical trial is to establish a predictive model for post-dural puncture headache,with the goal of implementing proactive interventions and treatments to reduce the incidence of PDPH and improve clinical management. Therefore, establishing an effective early warning model is crucial Participants will receive ultrasound, magnetic resonance imaging (MRI) and (or ) ICARE examinations before and after spinal puncture

ELIGIBILITY:
Inclusion Criteria:

BMI ≤ 30 kg/m² Normal liver and kidney function before surgery Normal coagulation function before surgery Hemoglobin > 70 g/L Platelet count > 80 × 10⁹/L

Exclusion Criteria:

Patients who experience major bleeding during or after surgery Patients with cerebrospinal fluid leakage or other serious malformations Patients with mental health disorders or cognitive dysfunction

Ages: 3 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients who need dural puncture
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (ONSD) measurement by MRI | 1 hour before dural puncture
  ONSD Measurement by MRI
Optic nerve sheath diameter (ONSD) measurement by MRI | 24 hours after dural puncture
  ONSD Measurement by MRI
Optic nerve sheath diameter (ONSD) measurement by B ultrasound | 1 hour before dural puncture
  ONSD Measurement by B ultrasound
Optic nerve sheath diameter (ONSD) measurement by B ultrasound | 8 hours after dural puncture
  ONSD Measurement by B ultrasound
Optic nerve sheath diameter (ONSD) measurement by B ultrasound | 24 hours after dural puncture
  ONSD Measurement by B ultrasound
Optic nerve sheath diameter (ONSD) measurement by B ultrasound | 48 hours after dural Puncture
  ONSD Measurement by B ultrasound
Intraocular Pressure messurement | 1 Hour before dural Puncture
  Intraocular Pressure measurement by Icare
Intraocular Pressure messurement | 8 hours after dural puncture
  Intraocular Pressure measurement by Icare
Intraocular Pressure messurement | 24 hours after dural puncture
  Intraocular Pressure measurement by Icare
Intraocular Pressure messurement | 48 hours after dural puncture
  Intraocular Pressure measurement by Icare

SECONDARY OUTCOMES:
number of punctures | 24 hours after dural puncture
  number of punctures
type of puncture needle | 24 hours after dural puncture
  type of puncture needle
Onset time of postoperative headache and duration | 24 hours after dural puncture
  Onset time of postoperative headache" and "duration

CONTACTS AND LOCATIONS:
Overall Officials: Yilin Zhao, Principal Investigator — Huazhong Universty of Science and Technology
Locations (1):
- Tongji Hospital of Tongji Medical College of Huazhong Universtiy of Science and Technology, Wuhan, Hubei, China